CLINICAL TRIAL: NCT06251414
Title: Study on the Effect of Blood Flow Restriction Training Combined With IASTAM on Symptoms in Patients With Chronic Ankle Instability
Brief Title: Study on the Effect of Exercise Intervention Combined With Physical Therapy on Chronic Ankle Instability Symptoms
Acronym: CAI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yang Liu (Other)
Responsible Party: Sponsor-Investigator, Yang Liu, doctor, Wuhan Sports University
Organization: Wuhan Sports University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Wuhan Sport University
Record Dates: First submitted 2024-01-08; First posted 2024-02-09 (Actual); Last update posted 2024-02-09 (Actual); Status verified 2024-02

CONDITIONS: Chronic Ankle Instability,CA
Keywords: Chronic Ankle Instability,CAI; Blood Flow Restriction Training，BFRT; Instrument-Assisted Soft Tissue Mobilization，IASTM; Tuina Massage
MeSH Terms: interventions — amobarbital, secobarital drug combination; Massage

STUDY DESIGN:
Intervention Model Description: There is no specific relevant model to refer to for use.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Blood Flow Restriction Training，BFRT (Experimental): Blood Flow Restriction Training (BFRT) is a special training technique aimed at limiting blood flow by using cuffs or elastic bands on the limbs to promote muscle growth and improve strength. BFRT was originally designed for rehabilitation injured athletes as it can improve muscle strength while reducing load, helping to avoid further injuries during the rehabilitation process. But as research deepens, it is gradually being applied to a wider range of fitness and training fields. One major advantage of BFRT is that it allows for efficient training under relatively light loads, reducing the burden on joints and tendons, making it suitable for people who find it difficult to withstand high-intensity training due to injuries or other reasons. Meanwhile, BFRT also has the characteristic of achieving muscle growth and strength growth in a short period of time, and it is considered a time-saving training method. BFRT can not only be used for strength training, but also for rehabilitation, i
  Interventions: Behavioral: Exercise Intervention
- Instrument-Assisted Soft Tissue Mobilization，IASTM (Experimental): Instrument Assisted Soft Tissue Mobilization (IASTM) is a physical therapy technique that utilizes specially designed tools (such as metal or plastic scraping boards) to assist in the treatment of soft tissue problems. Mainly used in rehabilitation medicine, sports medicine, and plastic surgery, it is used to handle tension, adhesion, pain, and motor dysfunction of muscles, fascia, and tendons. The edge design of IASTM special tools can loosen adhesions in tissues, improving their elasticity and plasticity. Regulating pathological areas through neural pathways, reducing pain and improving neurological function. And different types of treatment tools improve the accuracy of treatment, promote blood circulation, accelerate the rehabilitation process, improve tissue elasticity, expand joint range of motion, and have lower risks and complications compared to invasive surgery.
  Interventions: Behavioral: Instrument-Assisted Soft Tissue Mobilization
- Tuinal (Placebo Comparator): Tuinal is an important physical therapy method in traditional Chinese medicine, which can be traced back to the Shang Dynasty around 2700 BC. With the continuous development of social economy and cultural exchange, Tuinal technology based on traditional Chinese medicine ethics and guided by modern scientific theories gradually emerged. The technical treatment methods are mainly relaxation techniques, supplemented by movement techniques. Following the principle of combining movement and stillness, emphasizing both muscles and bones, and progressing step by step, massage has significant therapeutic effects on skeletal muscle diseases. In clinical practice, massage therapists use various techniques to apply to specific parts or acupoints of the human body, keeping the nerves and muscle tissues in a good state, improving the unblocking of meridians, relaxing soft tissues, restoring flexibility, and relieving symptoms such as muscle spasms and pain.
  Interventions: Behavioral: Tuinal

INTERVENTIONS:
Behavioral: Exercise Intervention — Blood Flow Restriction (BFR) training, also known as occlusion training or restricted blood flow training, involves applying external pressure to a limb using inflatable cuffs or elastic bands. This pressure partially restricts arterial blood flow while occluding venous blood flow in the pressured limb. The goal is to increase muscle strength and size by creating metabolic stress and promoting physiological adaptations, such as muscle hypertrophy, with lighter loads than traditional resistance training.
  Other Names: Blood Flow Restriction Training，BFRT
  Arms: Blood Flow Restriction Training，BFRT
Behavioral: Instrument-Assisted Soft Tissue Mobilization — Instrument-Assisted Soft Tissue Mobilization (IASTM) is a therapeutic technique that involves the use of specially designed tools or instruments to apply controlled mechanical pressure to soft tissues in the body. These tools are typically made of stainless steel or other materials and have various shapes and edges. The primary aim of IASTM is to address musculoskeletal conditions by breaking down scar tissue, fascial restrictions, and adhesions in the soft tissues. Practitioners use the instruments to detect and treat areas of tissue dysfunction, promoting improved range of motion, reduced pain, and enhanced functional mobility.
  Other Names: IASTM
  Arms: Instrument-Assisted Soft Tissue Mobilization，IASTM
Behavioral: Tuinal — Tuinal, also known as Tui Na or Chinese therapeutic massage, is a traditional Chinese medicine (TCM) healing technique that involves manual manipulation of the body's soft tissues, including muscles and tendons. It is a form of bodywork that aims to balance the flow of vital energy (Qi) within the body and promote overall well-being. Tuina techniques may include kneading, rolling, pressing, and brushing, and they are applied to specific acupressure points or along the body's meridians. Tuina is used to address various health concerns, alleviate pain, improve circulation, and enhance the body's natural healing processes, making it an integral part of traditional Chinese medicine.
  Other Names: massage
  Arms: Tuinal

SUMMARY:
Purpose; Through experimental observation of exercise intervention (blood flow restriction training combined with low load ankle muscle strength training and balance training) combined with instrument tool therapy (Instrument Soft Tissue Release Technique, IASTM), the intervention effect on ankle function, strength, and joint range of motion of sports dance athletes with ankle instability was observed.

Method; 45 subjects with unstable, restricted or uncomfortable ankle joints were selected as observation subjects and randomly divided into ankle blood flow restriction training combined with IASTM group (n=15), ankle blood flow restriction training alone (n=15), and traditional ankle strength training (n=15). The intervention lasted for 6 weeks, once a week. Cumberland ankle instability assessment, FAAM ankle function assessment score, and ankle range of motion measurement were performed at three time points before intervention, after the first intervention, and after 6 weeks of intervention for three groups. The ankle strength test was only compared and analyzed at two time points before and after intervention.

ELIGIBILITY:
Inclusion Criteria:

* Age: 18-35 years old
* Course of illness: Suffering from chronic ankle instability symptoms that last for at least 3 months
* Symptoms: Ankle instability, frequent ankle sprains, discomfort during walking or exercise
* Functional screening: Two or more tests tested positive for ankle joint function screening before the experiment
* Structural examination: No joint structural lesions or congenital ankle deformities,
* Medical history: Have not undergone ankle surgery or have external injuries
* Health status: No serious heart, lung, nervous system or other systemic diseases
* Exercise level: Able to complete the exercise intervention and evaluation tasks specified in the experiment
* Agree to participate in the study: Has limited exercise ability and is unable to complete the research task

Exclusion Criteria:

* Under 18 years old or over 35 years old
* Acute ankle injury or no joint injury
* No ankle instability or unwillingness to cooperate with research requirements
* Failed ankle function screening
* Structural lesions or congenital ankle deformities present in the ankle joint
* Have undergone ankle surgery or have obvious injuries or wounds
* Serious heart, lung, nervous system or other systemic diseases
* Due to limited athletic ability, unable to complete research tasks
* Disagree to participate in the study, or inability to understand and comply with the research protocol

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 45 (Actual)
Dates: Start 2023-11-20 (Actual); Primary Completion 2023-11-30 (Actual); Study Completion 2023-12-30 (Actual)

PRIMARY OUTCOMES:
Cumberland Ankle Instability Tool，CAIT | 4-6week
  Evaluated the patient's perception of ankle instability, including the frequency, CAIT typically includes a specific range of questions, each of which may have different scores. The total score is usually between 0 and 30 points, with higher scores indicating higher stability intensity, and impact of symptoms
Foot and Ankle Ability Measure（FAAM） | 4-6week
  Foot and Ankle Ability Measure (FAAM) is a scale used to evaluate ankle joint function, which includes questions about pain, function, and quality of life, and can be used to assess the overall condition of patients with ankle instability. The functional score includes two types of assessments: the functional level of daily life (FAAM-ADL) and the functional level of physical activity (FAAM-SPORT). The score range is usually from 0 to 100, where 100 represents completely normal ankle joint function, and 0 represents extreme restriction or complete inability to use the ankle joint.
Ankle joint range of motion | 4-6week
  This study used a high-precision joint motion angle measuring ruler to measure the range of motion of different ankle functions in both sitting and supine positions, including measurements of dorsiflexion and plantar flexion of the ankle, as well as measurements of varus and eversion of the foot. The larger the angle, the better the improvement in joint motion.
Ankle joint strength test | 4-6week
  The experimental strength data was tested using a handheld digital muscle strength tester (model: FM-204M series muscle strength tester). The measurement unit of this muscle strength tester is N, with a measurement unit range of ± 50kgf and a measurement accuracy of ± 0.5% FS (range) ± 1 digital peak. The measured data includes both peak strength and instantaneous strength values. Therefore, this study used a handheld digital muscle strength tester, where participants sat in a suitable position, fixed the bottom of the instrument on the ground, and then applied force in different directions through their ankles. Measure the maximum force in the direction of dorsiflexion and plantarflexion of the ankle joint, abduction and eversion of the foot, and adduction and eversion. The strength test for each different exercise segment needs to be completed three times, and the average of the maximum strength values from the three tests is taken.

CONTACTS AND LOCATIONS:
Locations (1):
- YangLiu, Wuhan, Hubei, China

IPD SHARING:
Plan to Share IPD: No
This study requires me to conduct more experimental verification.

REFERENCES:
- [Derived] Liu Y, Wang Y. Study on the effect of blood flow restriction training combined with IASTAM on ankle strength and function intervention in athletes with chronic ankle instability in sport dance events. BMC Sports Sci Med Rehabil. 2024 Apr 11;16(1):81. doi: 10.1186/s13102-024-00873-x. PMID 38605396

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-12-30): https://cdn.clinicaltrials.gov/large-docs/14/NCT06251414/Prot_SAP_000.pdf
  • Informed Consent Form (2023-12-30): https://cdn.clinicaltrials.gov/large-docs/14/NCT06251414/ICF_001.pdf